CLINICAL TRIAL: NCT04505930
Title: Developing and Pilot Testing a Multilevel HPV Vaccination Intervention in Chinese American Community
Brief Title: Pilot HPV Vaccination in Chinese American Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pilot HPV Vaccination; U54CA153513 (NIH)
Record Dates: First submitted 2020-07-23; First posted 2020-08-10 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: HPV

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group with active education (Experimental): The study team provides participants in the intervention group with interventional education, using interactive video watch and dynamic discussion.
  Interventions: Behavioral: Interventional HPV vaccination video modules
- Control Group with handouts (Active Comparator): The study team provides the participants in the control group with education, using only handouts of vaccinations including HPV, but not using interactive video watch and dynamic discussion
  Interventions: Behavioral: General Vaccination Education

INTERVENTIONS:
Behavioral: Interventional HPV vaccination video modules — The study team provide participants in the intervention group with interventional education, using interactive video watch and dynamic discussion. The educational videos were aiming to reinforcement and improvement the awareness, knowledge, attitude, intention and actual uptake of HPV vaccination shots among Chinese parents.
  Arms: Intervention Group with active education
Behavioral: General Vaccination Education — Education session conducted using only handouts of vaccinations including HPV
  Arms: Control Group with handouts

SUMMARY:
This study provides a pioneer model in increasing knowledge of HPV vaccination among Chinese American families through culturally tailored interventions, and eventually increase the HPV vaccine uptake among Chinese American adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified Chinese Parents or legal guardian with children aged 11-18 years old;
2. The children have not received any does of HPV vaccination

Exclusion Criteria:

-

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
changes from baseline HPV vaccine uptake rate at 6-month follow up | baseline, and 6-month follow up
  the rate of getting HPV vaccination uptake 6 months post intervention

SECONDARY OUTCOMES:
change of HPV knowledge from baseline to 6-month follow up | baseline, and 6-month
  Knowledge scores ranged from 0 to 7, computed by taking the total number of correct answers to the questions with a higher numeric value indicating better knowledge
change in adolescents engagement percentage | baseline, and 6-month
  change in the percents of engaging adolescents in decision-making at post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Grace X Ma, PhD, Principal Investigator — Temple University
Locations (1):
- Center for Asian Health, Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania, United States